CLINICAL TRIAL: NCT04674059
Title: A Descriptive Study on Patients With Bipolar Disorder in Rwanda
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Collaborators: University of Rwanda (Other); Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AUUR2020DKRW_3
Record Dates: First submitted 2020-12-04; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Mental Disorder; Bipolar Disorder
MeSH Terms: conditions — Mental Disorders; Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: patient survey — A questionnaire will be delivered by the health care providers at Ndera Hospital, Kigali, Rwanda or CHUK, Hospital, Kigali, Rwanda. The questions will explore the patient's clinical characteristics, the current treatment and their experience with the mental health care system.

SUMMARY:
The aim is to provide a comprehensive assessment regarding the service provision and the accessibility to intensive mental health care in Rwanda

DETAILED DESCRIPTION:
The aim is to provide a comprehensive assessment regarding the service provision and the accessibility to intensive mental health care in Rwanda for patients with bipolar disorder.

Knowing about the barriers to treatment, risk and protective factors as well as the current treatment offered for patients with bipolar disorder is essential for the development of therapeutic approaches and improvement in access to care. Up to now, no data on characteristics of patients with bipolar disorder in Rwanda and related risk and protective factors is available. For this purpose, all outpatients with bipolar disorder in Rwanda age > 18 years, will over a 1-year period be invited to participate in a survey on their experience living with bipolar disorder in Rwanda. Moreover, patients and relatives will be invited for in-depth interviews to explore their perceptions and experiences with the mental health system. Health care providers will meet for focus discussions on to assess the experience, knowledge and practice of caregiving for individuals with bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Bipolar Disorder type I or II that meets DSM-V diagnostic criteria
* Age ≥ 18 years

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Outpatients with bipolar disorder in Rwanda
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnoses | 1 year
  Psychiatric diagnoses including both primary diagnosis, secondary diagnosis and somatic comorbidity.
Diagnostic delay | 1 year
  Age of individual at onset of symptoms and age when diagnosed with bipolar disorder.
Number of previous psychiatric hospitalisations | 1 year
  Numerical value of the previous psychiatric hospitalisations.
Number of previous crises | 1 year
  Numerical value of the previous crises defined as an episode of depression or mania or hypomania.
Types of medical treatment provided | 1 year
  What type of medical treatment is provided, including brand name, administration and dosage.
Medical Adherence | 1 year
  Medication Adherence Rating Scale (MARS) will be used to assess beliefs and barriers to medication adherence. Total scores on the MARS may range between 0 and 10, with a higher score indicating better medication adherence.
The referral pathways | 1 year
  Who initiated the first contact, who did you seek for help, what kind of help was provided, percent of patients who came in contact with traditional leaders.
Degree of internal stigma | 1 year
  Internalized Stigma of Mental Illness Inventory - 9-item Version (ISMI-9) will be used to assess self-stigma. The resulting score should range from 1 to 4. A score ranging between 1.00-2.50: does not report high internalized stigma vs. a score ranging between 2.51-4.00: indicating high internalized stigma.

CONTACTS AND LOCATIONS:
Overall Officials: Per Kallestrup, Prof., Study Chair — University of Aarhus

IPD SHARING:
Plan to Share IPD: No